CLINICAL TRIAL: NCT00456040
Title: Characteristics of Patients With Systemic Amyloidosis and Severe Heart Failure Being Evaluated for a Sequential Cardiac and Autologous Stem Cell Transplantation
Brief Title: Characteristics of Patients With Amyloidosis & Heart Failure Being Evaluated for a Heart Transplant
Status: Completed | Type: Observational
Sponsor: Massachusetts General Hospital (Other)
Other Study IDs: 2007-p-000302
Record Dates: First submitted 2007-04-02; First posted 2007-04-04 (Estimated); Last update posted 2007-04-04 (Estimated); Status verified 2007-04

CONDITIONS: Cardiomyopathy
Keywords: amyloidosis; heart failure; heart transplant; stem cell transplant
MeSH Terms: conditions — Cardiomyopathies; Amyloidosis; Heart Failure

STUDY DESIGN:
Observational Model: Defined Population | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

SUMMARY:
The purpose of this study is to describe the characteristics of patients with amyloidosis and severe heart failure being evaluated for cardiac and stem cell transplantation.

DETAILED DESCRIPTION:
Systemic amyloidosis is a progressive disease leading to organ failure and death. Treatment has improved survival with stem-cell transplantation. Unfortunately, patients with amyloidosis and severe heart failure are not eligible for stem-cell transplantation.

The average rate of survival for patients with amyloidosis who receive a heart transplant is decreased.

Previous trials have raised the possibility that survival may be increased in patients with amyloidosis, if chemotherapy and stem-cell transplantation is performed after a heart transplant.

We plan to review data of patients with amyloidosis and heart failure who were being evaluated for a heart transplant.

ELIGIBILITY:
Inclusion Criteria:

* Patients with amyloidosis
* NYHA class III or IV heart failure
* Patients undergoing heart transplant evaluation
* Patients less than 18 years of age

Exclusion Criteria:

* Patients who have unstable pulse and blood pressure

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25
Dates: Start 2007-03; Study Completion 2007-03

CONTACTS AND LOCATIONS:
Overall Officials: Marc J Semigran, MD, Principal Investigator — Massachusetts General Hospital